CLINICAL TRIAL: NCT04410926
Title: Clinical And Radiological Outcomes Of Corrective Exercises With Neuromuscular Electrical Stimulation In Children And Flexible Flatfeet: A Randomized Controlled Trial
Brief Title: Corrective Exercises With Neuromuscular Electrical Stimulation In Children With Flexible Flatfeet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Mahmoud Abd-elmonem, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Children With Flatfeet
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Sports Physical Therapy
Keywords: Foot arch; Foot print; Idiopathic flexible flatfoot; Navicular height; Short foot exercises.

STUDY DESIGN:
Intervention Model Description: Intervention:
  Corrective exercises The experimental and control groups performed a designed strengthening exercises included short-foot exercise, toes-spread-out exercise, toes-extension exercise and toe-curls for 60 minutes. Each exercise was performed for 30 repetitions holding each repetition for 5 seconds (about three minutes).
  Neuromuscular electrical stimulation The experimental group received NMES aiming to reinforce the planter intrinsic foot muscles. The surface electrodes were placed over the abductor halluces based on the evidence that it has the largest cross-sectional area of the intrinsic foot muscles
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): Corrective exercises The experimental and control groups performed a designed strengthening exercises included short-foot exercise, toes-spread-out exercise, toes-extension exercise and toe-curls for 60 minutes. Each exercise was performed for 30 repetitions holding each repetition for 5 seconds (about three minutes).
  Neuromuscular electrical stimulation The control group received placebo NMES with no current stimulation. In another words, the current intensity was set at 0mA while standing on both feet for 30 minutes.
  Interventions: Other: Corrective exercises
- intervention group (Experimental): Corrective exercises The experimental and control groups performed a designed strengthening exercises included short-foot exercise, toes-spread-out exercise, toes-extension exercise and toe-curls for 60 minutes. Each exercise was performed for 30 repetitions holding each repetition for 5 seconds (about three minutes).
  Neuromuscular electrical stimulation
  The experimental group received NMES aiming to reinforce the planter intrinsic foot muscles. High-voltage pulsed current was set at frequency of 85 Hz with 5 seconds contraction time and 12 seconds rest time while the ramp-up and ramp-down time were 0.3 and 0.7 respectively. The current intensity was adjusted based on the individual tolerance without reporting pain or discomfort while standing on both feet. The stimulation time lasted each session for 30 minutes.
  Interventions: Other: Corrective exercises; Other: Neuromuscular electrical stimulation

INTERVENTIONS:
Other: Corrective exercises — The experimental and control groups performed a designed strengthening exercises included short-foot exercise, toes-spread-out exercise, toes-extension exercise and toe-curls for 60 minutes
Other: Neuromuscular electrical stimulation — The experimental group received NMES aiming to reinforce the planter intrinsic foot muscles for 30 minutes. The surface electrodes were placed over the abductor halluces. The control group received placebo NMES with no current stimulation.
  Arms: intervention group

SUMMARY:
flexible flatfoot is a common foot misalignment in children. various treatment procedures are used to correct or to avoid future complain among adults and pediatric population.

DETAILED DESCRIPTION:
Ethics Statement This study was approved by the Institutional Review Board of the Faculty of Physical Therapy, Cairo University, Egypt (no. P.T.REC/012/0016370) and strictly adhered to the criteria proclaimed in the latest version of the Declaration of Helsinki code of ethics. Children's participation was commissioned by asking their legal guardian to sign a consent form prior to data collection.

Study design A prospective double-masked randomized controlled trial was carried out from September 1, 2018 to December 31, 2019 at the Out-patient Physical Therapy Clinic of Faculty of Physical Therapy, Cairo University.

Sample size estimation Sample size calculation was performed prior to the study using G*POWER statistical software (version 3.1.9.2; Franz Faul, Universitat Kiel, Germany) [F tests- MANOVA. Estimates of means of SAI were calculated from a preliminary study included 10 children who were assigned to the two treatment groups (5 children for each). Repeated measures, within-between interaction, α=0.05, β=0.2, Pillai V = 0.1, and large effect size] and revealed that the appropriate sample size for this study was not less than 65 children. ¬then, 70 children were recruited to account for the possible dropout rates.

Randomization Seventy-two volunteer children who were recruited from governmental schools at Cairo and Giza Provinces. The online Graph Pad software was used to allocate study participants to either intervention group (corrective exercise and NMES) control group (corrective exercise and placebo NMES). All children/legal and examiners were unaware of group allocation.

ELIGIBILITY:
Inclusion Criteria:

The criteria for inclusion were

* Di¬agnosed (by an orthopedist) with asymptomatic FFF,
* Navicular height more than 9-millimeter (mm),
* Grade III flatfoot grade (midfoot width exceeding forefoot width)
* Normal body weight (BMI from 5th to 85th percentile),
* Presented with no neuromuscular or osseous anomalies.

Exclusion Criteria:

The authors excluded all children who had a history of

* Symptomatic flatfeet
* Congenital deformities of the lower extremities (e.g. genu valgum, femoral anteversion, leg length discrepancy, hypermobile joint)
* Scar/irri¬tated skin at the electrode placement
* Neurological/ neuromuscular disorders.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Staheli's arch index | period of the treatment was 4 successive months
  The footprint is one of the easy, cost effective, noninvasive and objective measures for assessing the SAI. A value of SAI >1.15 indicates flatfeet.
Navicular height | period of the treatment was4 successive months
  The navicular height was measured by the navicular drop test first described by Brody21 to evaluate the amount of foot pronation. Measurements of 6-9 mm are considered to be within the normal range. It represents the vertical extension between the most prominent point of the navicular and the supporting surface.
Radiographic indexes | period of the treatment was 4 successive months
  Radiographic indexes were carried out through bilateral radiographs encompassing horizontal (antero-posterior) and sagittal (lateral) views obtained with the child in a relaxed bipedal weight-bearing erect standing.

CONTACTS AND LOCATIONS:
Overall Officials: Emam H El-Negamy, Study Chair — Cairo University; Mahmoud A Mahran, Study Director — Ain Shams University, Egypt; Asmaa T Ramadan, Principal Investigator — Cairo university, Egypt
Locations (1):
- faculty of physical therapy, Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Evans AM, Rome K, Carroll M, Hawke F. Foot orthoses for treating paediatric flat feet. Cochrane Database Syst Rev. 2022 Jan 26;1(1):CD006311. doi: 10.1002/14651858.CD006311.pub4. PMID 35080267
- [Derived] Evans AM, Rome K, Carroll M, Hawke F. Foot orthoses for treating paediatric flat feet. Cochrane Database Syst Rev. 2022 Jan 14;1(1):CD006311. doi: 10.1002/14651858.CD006311.pub3. PMID 35029841